CLINICAL TRIAL: NCT04095195
Title: Italian Registry of Families At Risk of Pancreatic Cancer
Brief Title: Registry of Subjects at Risk of Pancreatic Cancer
Acronym: IRFARPC
Status: Recruiting | Type: Observational
Sponsor: Associazione Italiana per lo Studio del Pancreas (Other)
Responsible Party: Sponsor
Other Study IDs: IRFARPC
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Familial Pancreatic Cancer; BRCA1 Mutation; BRCA2 Mutation; Lynch Syndrome; FAMMM - Familial Atypical Mole Malignant Melanoma Syndrome; Hereditary Pancreatitis; Peutz-Jeghers Syndrome
Keywords: Familial Pancreatic Cancer; BRCA Mutation; Lynch Syndrome; Screening pancreatic cancer; Surveillance pancreatic cancer
MeSH Terms: conditions — Pancreatic carcinoma, familial; Colorectal Neoplasms, Hereditary Nonpolyposis; Dysplastic Nevus Syndrome; Hereditary pancreatitis; Peutz-Jeghers Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Familial pancreatic cancer relatives
  Interventions: Radiation: MRCP; Procedure: Endoultrasonography
- Peutz-Jeghers syndrome
  Interventions: Radiation: MRCP; Procedure: Endoultrasonography
- BRCA 1/2, PALB2, p16 mutations with familiarity for PC: Known genetic mutation and at least 1 1st- or 2nd-degree relative suffering from PC
  Interventions: Radiation: MRCP; Procedure: Endoultrasonography
- Lynch syndrome with familiarity for pancreatic cancer
  Interventions: Radiation: MRCP; Procedure: Endoultrasonography
- FAMMM syndrome
  Interventions: Radiation: MRCP; Procedure: Endoultrasonography
- Hereditary and genetic pancreatitis
  Interventions: Radiation: MRCP; Procedure: Endoultrasonography

INTERVENTIONS:
Radiation: MRCP — Subjects fulfilling the "radiological follow-up criteria" will be submitted to MRCP or EUS according to the pancreatologist's prescription
Procedure: Endoultrasonography — Subjects fulfilling the "radiological follow-up criteria" will be submitted to MRCP or EUS according to the pancreatologist's prescription

SUMMARY:
IRFARPC is a multicenter national registry designed to study the diagnosis and predisposing factors of subjects with an inherited increased risk for pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is a devastating disease with a dismal prognosis. One of the ways to improve survival might be early detection.

Within years, many predisposing diseases or genetic conditions have been identified, thus screening/surveillance have been established worldwide.

A registry of subjects at risk of pancreatic cancer will has been built up to investigate the possibility of diagnosis pancreatic cancer, or one if its predisposing lesions.

Inclusion criteria will be adopted as "enrollment criteria". According to this, individuals > 18 years old will be enrolled; their familiar history and/or genetic predisposition will be collected, as well as current or previous medical records/medications data. Thereafter, according to specific age-based criteria, those individuals initially enrolled will be will be considered for a "surveillance protocol" ("interventional follow-up criteria") and they will be submitted to Cholangio-Wirsung Magnetic Resonance or Pancreatic Endoultrasonography according to the pancreatologist's prescription at each participating center.

Individuals suffering from the following conditions will be enrolled:

familial pancreatic cancer; Peutz-Jeghers syndrome; a known BRCA-2, BRCA-1, PALB2, or p16 mutation with at least one first- or second-degree relative suffering from pancreatic cancer; hereditary pancreatitis; FAMMM syndrome; Lynch syndrome with at least one first- or second-degree relative suffering from pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria to enter the registry:

* individuals with at least two relatives suffering from pancreatic cancer, with at least 1 first-degree and until the third-degree
* subjects with known genetic mutation of BRCA2, BRCA1, p16, PALB2 with at least 1 first- or 2nd-degree relative suffering from pancreatic cancer
* subjects suffering from FAMMM Syndrome
* subjects suffering from Peutz-Jeghers Syndrome
* subjects suffering from PRSS-1- or CFTR- or SPINK-1- related pancreatitis
* subjects suffering from Lynch syndrome with at least 1 first- or 2nd-degree relative suffering from pancreatic cancer

Inclusion criteria to join the "radiologic follow-up":

* 45 years or 10 years younger than the youngest index case of pancreatic cancer in the family for familial cases
* 40 years or 5 years younger than the youngest index case of pancreatic cancer for subjects suffering from hereditary/genetic pancreatitis, Lynch syndrome, or carrying a known BRCA 1/2, PALB2, p16 genetic mutation with familiarity for pancreatic cancer
* 30 years for subjects suffering from FAMMM, Peutz-Jeghers syndrome

Exclusion Criteria:

- pregnancy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects at high-risk of pancreatic cancer will be enrolled and a surveillance examination will be performed according to inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2044-08-20 (Estimated); Study Completion 2045-09-20 (Estimated)

PRIMARY OUTCOMES:
This clinical study will assess the diagnostic yield of a clinical surveillance program for pancreatic neoplasia or predisposing conditions (PanIN, IPMNs) in high risk individuals | 25 years
  Number of malignant and pre-malignant lesions diagnosed over time

SECONDARY OUTCOMES:
This study will investigate possible risk factors for the incidence or the progression of for pancreatic neoplasia or predisposing conditions (PanIN, IPMNs) in high risk individuals | 25 years
  Identification of risk factors for malignant or pre-malignant lesions diagnosis

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Ospedale Pederzoli, Peschiera del Garda, Verona
  - San Raffele Vita Salute University Hospital, Milan
  - Chirurgia Generale e del Pancreas, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paiella S, Capurso G, Cavestro GM, Butturini G, Pezzilli R, Salvia R, Signoretti M, Crippa S, Carrara S, Frigerio I, Bassi C, Falconi M, Iannicelli E, Giardino A, Mannucci A, Laghi A, Laghi L, Frulloni L, Zerbi A. Results of First-Round of Surveillance in Individuals at High-Risk of Pancreatic Cancer from the AISP (Italian Association for the Study of the Pancreas) Registry. Am J Gastroenterol. 2019 Apr;114(4):665-670. doi: 10.1038/s41395-018-0414-z. PMID 30538291
- [Derived] Paiella S, Capurso G, Carrara S, Secchettin E, Casciani F, Frigerio I, Zerbi A, Archibugi L, Bonifacio C, Malleo G, Cavestro GM, Barile M, Larghi A, Assisi D, Fantin A, Milanetto AC, Fabbri C, Casadei R, Donato G, Sassatelli R, De Marchi G, Di Matteo FM, Arcangeli V, Panzuto F, Puzzono M, Dal Buono A, Pezzilli R, Salvia R, Rizzatti G, Casadio M, Franco M, Butturini G, Pasquali C, Coluccio C, Ricci C, Cicchese N, Sereni G, de Pretis N, Stigliano S, Rudnas B, Marasco M, Lionetto G, Arcidiacono PG, Terrin M, Crovetto A, Mannucci A, Laghi L, Bassi C, Falconi M. Outcomes of a 3-Year Prospective Surveillance in Individuals at High Risk of Pancreatic Cancer. Am J Gastroenterol. 2024 Apr 1;119(4):739-747. doi: 10.14309/ajg.0000000000002546. Epub 2023 Oct 3. PMID 37787643